CLINICAL TRIAL: NCT06471790
Title: Movement Observation and Tracking In Obstetrics - Epidural and Ambulation Feasibility Study Using Inertial Sensors
Brief Title: Inertial Sensors for Obstetrical Walking Epidural Tracking
Acronym: MOTION-EASE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0097; 2024-A00279-38 (Other: ID-RCB)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related; Epidural; Anesthesia, Headache; Labor Complication
Keywords: PREGNANCY; LABOR; EPIDURAL ANALGESIA; WALKING EPIDURAL; MOVEMENTS; GAIT; INERTIAL SENSOR
MeSH Terms: conditions — Headache; Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Walking Epidural Analgesia for Labor: Pregnant women in labor who benefit from walking epidural analgesia technique will be monitored using inertial wearable sensors beginning from the first stage of labor and up to delivery.

SUMMARY:
Freedom of movement and the ability to walk are crucial during the first stage of labor, potentially reducing labor duration, cesarean section risk, epidural analgesia use, and bladder catheterization. While the clinical effects of ambulation during labor remain controversial, there is a consensus on its positive impact on the birthing experience and satisfaction.

Epidural analgesia remains the gold standard for pain control during labor, with a utilization rate of 82% in France. Recent advancements in obstetric analgesia have allowed for lower doses of analgesics, often administered via patient-controlled analgesia, which maintains the potential for ambulation during labor. However, only a small number of maternity units in France offer this technique. The main barriers include organizational issues such as unsuitable facilities, lack of wireless telemetry, and potential risks such as falls and hypotension.

Significant changes in gait characteristics are observed throughout pregnancy, particularly during the third trimester, and are studied in laboratory settings using video capture and analysis. Gait during labor is influenced by pain, fetal progression, and anatomical changes in the pelvis. The presence of epidural analgesia, where local anesthetics likely affect neural transmission, may impact motor commands and sensory feedback, further altering gait characteristics. These biomechanical aspects of labor remain understudied.

Wearable inertial sensors show promise in maternal health monitoring by providing real-time data for motion and gait studies. However, their application has not been described or validated during labor, particularly in walking conditions. Continuous dynamic study of gait in these conditions could enable non-invasive, non-intrusive monitoring of analgesia effectiveness, fall risk prediction, and labor progression analysis.

The aim of this feasibility study is to validate the use of wearable inertial sensors to quantify movements and characterize gait during the first stage of labor, both with and without low-dose epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy >= 38 gestation weeks
* no significant medical history (American Society of Anesthesiologists class ASA 1)
* receiving low-dose epidural analgesia with ambulation (in accordance with current service protocol)
* not opposed to the study

Exclusion Criteria:

* Refusal to participate in this study
* Non-French-speaking patient
* History of osteoarticular pathology likely to change gate (severe scoliosis, spinal surgery, congenital hip deformity, pelvic fracture, ligament or knee joint pathology)
* adults under legal protection
* multiple pregnancy
* need for continuous intravenous infusion with infusion stand during ambulation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: at-term (>= 38 gestation weeks) women admitted to the maternity facility for labor and delivery and willing low dose epidural analgesia with walking option
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-07-12 (Estimated); Study Completion 2026-07-12 (Estimated)

PRIMARY OUTCOMES:
triaxial (x, y, z) velocity changes over time unit (dV/dt) = m/s2 (meter over square second) | during walking starting from the demand of the parturient to have an epidural up to delivery
  gait patterns derived from accelerometer data measuring acceleration in three axes (x, y, z)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail PH DZIADZKO, MD, Principal Investigator — Anesthésie Réanimation Douleur
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No